CLINICAL TRIAL: NCT05926245
Title: Topical Absorption of Glutathione-cyclodextrin Complex in Healthy Human Subjects Improves Immune Response Against Mycobacterium Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Ali Badaoui, Osteopathic Medical Student, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: antioxidants-2402271
Record Dates: First submitted 2023-06-17; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Glutathione-cyclodextrin Complex Absorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): 15 adult healthy volunteers to serve as controls for the experimental group. This group will receive a placebo-topical spray with empty nanoparticles.
  Interventions: Dietary Supplement: Placebo Solution
- Glutathione Group (Experimental): 15 adult healthy volunteers will serve in the experimental group. This group will receive glutaryl treatment topical spray with nanoparticles containing GSH.
  Interventions: Dietary Supplement: Glutaryl Solution

INTERVENTIONS:
Dietary Supplement: Glutaryl Solution — Glutathione, ascorbic acid, cyclodextrin, potassium sorbate and radish root extracts
  Arms: Glutathione Group
Dietary Supplement: Placebo Solution — Empty nanoparticles
  Arms: Placebo Group

SUMMARY:
The proposed clinical trial will confirm the therapeutic absorption of glutathione following topical Glutaryl application in increasing blood GSH levels without an invasive procedure.

GOAL: Confirm therapeutic level of glutathione following topical transdermal application.

HYPOTHESIS: The hypothesis of the proposed study is that the glutathione administration will increase RBC levels of glutathione above 80%.

AIM: Determine a non-invasive way to increase glutathione levels in the plasma and blood cells.

This aim will be accomplished as follows:

STEP 1: We will recruit eligible healthy participants in the two study groups who are not currently taking any glutathione or N-acetyl cysteine (NAC) supplementation.

STEP 2: Determine baseline levels of GSH, free radicals and cytokines through analysis of venipuncture blood draws.

STEP 3: Study subjects will be asked to spray themselves with either placebo or Glutaryl four times twice a day for three days on the ventral part of the abdomen. Measure the levels of GSH, free radicals and cytokines after 1 hour, 4 hour and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Control group) will include 15 healthy volunteers with the age group between 21-65. Participants belonging to Group 1 will be recruited from the local area. Group 1 will serve as controls for Group 2.

Group 2 (Glutathione Group) will include 15 healthy volunteers that are not allergic to any components of GlutarylTM who will be sprayed four times twice a day for three days with Topical glutathione Complex (GlutarylTM) formulation on their skin on their ventral part of the abdomen.

Components of Glutaryl:

Main ingredients of Glutaryl are Glutathione, ascorbic acid and cyclodextrin. The preservative system used is potassium sorbate and radish root extracts.

Exclusion Criteria:

* Pregnant and breastfeeding women. Anyone below age of 21 or above age of 65. Patients with active cancer. Patients with known liver disease, hepatitis, COVD-19, HIV, or AIDS. Patients taking some form of glutathione. Subjects who have previously fainted following venipuncture will also be excluded. By interviewing the subjects we will determine whether or not the subject will be excluded from the study based on their previous phlebotomy experiences.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
GSH | 72 hours
  Levels of total, reduced, and oxidized forms of GSH in the isolated plasma, red blood cells (RBCs) and peripheral blood mononuclear cells (PBMCs) isolated from the peripheral blood of the two-study groups will be assayed by spectrophotometry using an assay kit from Arbor Assays (3-12).

SECONDARY OUTCOMES:
Free Radicals | 72 hours
  To demonstrate that increased levels of GSH in the experimental group is accompanied by decreased levels of reactive oxygen species (ROS), free radical activity will be measured by malondialdehyde (MDA) assay that measures several end products of lipid peroxidation (3-12).
Pro- and Anti-inflammatory Cytokines | 72 hours
  To demonstrate that increased levels of GSH in the experimental group is accompanied by altered levels of pro- and anti-inflammatory cytokines and chemokines, we will measure the levels of pro- and anti-inflammatory cytokines and cytokines in the plasma derived from the two study groups by ELISA using an assay kit from ThermoFisher.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Ochoa, MD, Study Director — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT05926245/Prot_ICF_000.pdf